CLINICAL TRIAL: NCT03242798
Title: Assessment of Nutritional Status of Patients With Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: Harokopio University (Other)
Collaborators: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Meropi Kontogianni, Assistant Professor, Harokopio University
Other Study IDs: 105
Record Dates: First submitted 2017-08-02; First posted 2017-08-08 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Cirrhosis; Malnutrition
Keywords: liver cirrhosis; malnutrition; nutritional status; nutritional assessment
MeSH Terms: conditions — Fibrosis; Malnutrition; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cirrhosis is the twelfth leading cause of death worldwide. Malnutrition is prevalent among cirrhotic patients and is an important prognostic factor. Nutritional assessment is therefore crucial for identifying patients at risk or with already established malnutrition and refer them for nutritional intervention and support. In the current literature, nutritional assessment of cirrhotic patients is performed using several tools and methods. However their accuracy is widely affected by the underline disease and its complications. In addition, for the majority of the parameters under study, no gold standard tools and methods have been established so far. Studies on nutritional assessment in cirrhosis usually focus on one or few aspects of nutritional status and not on a full nutritional assessment combining information from medical, biochemical, nutritional, and body composition variables. Hence, the present study aims at a thorough assessment of the nutritional status of 170 cirrhotic patients using multiple widely available tools and methods, in order to assess their accuracy and estimate the prevalence of multiple malnutrition phenotypes such as undernutrition, sarcopenia, sarcopenic obesity and cachexia.

DETAILED DESCRIPTION:
The study sample will comprise of 170 adults with biopsy proven cirrhosis. A detailed medical and nutritional assessment will be implemented at baseline. For patients that will receive an intervention aiming at the cause of cirrhosis (e.g. antivirus therapy for HCV or HBV) the baseline assessment will take place before the beginning of the therapy and will be repeated three months after the completion of the medical intervention to explore the impact of the intervention on nutritional status. Data regarding the survival of all the patients will be collected one year after the baseline assessment.

More specifically regarding the detailed assessment, firstly, hepatologists of the research team will complete a full medical record regarding the primary disease, cirrhosis' complications, comorbidities and medication. The severity of cirrhosis will be assessed using the Child-Pugh score. Furthermore, in the Laboratory of Clinical Nutrition & Dietetics at Harokopio University, patients will participate in the following procedures:

* Anthropometry: Weight, height, waist and mid-arm circumference, and triceps skinfold will be measured. Body mass index, mid-arm muscle circumference and area will be estimated using standard equations.
* Body composition analysis: Total body DXA (Lunar DPX-MD, Madison, WI, USA) will be performed.
* Muscle strength and performance status: Handgrip strength measurement based on certain protocol and the "Short Physical Performance Battery" tool will be implemented.
* Dietary intake evaluation: Three non-consecutive 24h recalls (two weekdays and one weekend day) will be recorded. Data will be analyzed to estimate energy, macro- and micronutrients intake (Nutritionist Pro software, 2.2 version). Food group intake and meal patterns will also be evaluated.
* Physical activity assessment: Patients' physical activity levels will be assessed using the "Harokopio Physical Activity Questionnaire".

For patients with available upper abdomen computed tomographies skeletal muscle index at L3 will be calculated with the software SliceOmatic V5.0 software, Tomovision, Montreal, PQ. In addition, patients' nutritional risk or nutritional status will be assessed through several previously validated tools like the Subjective Global Assessment, the Royal Free Hospital Global assessment scheme and Liver Disease Undernutrition Screening Tool, the efficacy of which will be tested in the present study. Patients will be also categorized according to ESPEN's recent malnutrition diagnostic criteria.

The full assessment will be repeated only for patients who will receive an intervention aiming at the cause of cirrhosis (e.g. antivirus therapy for HCV or HBV) three months after the completion of the medical intervention.

One year after the baseline assessment of the study samples, data will be collected regarding survival, development of complications and decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Adults with biopsy proven cirrhosis.

Exclusion Criteria:

Patients with hepatocellular carcinoma, in hepatic coma, with acquired immunodeficiency syndrome, with renal or pancreatic insufficiency, receiving enteral nutrition or being pregnant, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will comprise of 170 adults with biopsy proven cirrhosis visiting hospital Liver Outpatient Clinics in Athens, Greece.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of malnutrition phenotypes. | Baseline
  Prevalence of different malnutrition phenotypes (e.g. undernutrition, sarcopenia, sarcopenic obesity), in cirrhotic patients of different disease stages, by implementing a thorough nutritional assessment.

SECONDARY OUTCOMES:
Survival. | One year after baseline measurements
  Assessment of survival one year after baseline measurements and association with the malnutrition phenotypes at baseline.
Validity test of available tools. | Baseline
  Test the sensitivity, specificity, positive and negative prognostic values of already available tools for nutritional screening or assessment against a combined index as the reference tool. If no tool is estimated as valid, a new combination of nutritional, biochemical and/or clinical parameters will be synthesized and its validity as a new screening or assessment tool will be assessed for the detection of cirrhotic patients at risk of malnutrition or already malnourished.
Nutritional status after medical treatment according to the etiology of cirrhosis. | 6 months after baseline measurements
  Changes in the nutritional status after medical treatment according to the etiology of cirrhosis, namely antivirus therapy for HCV or HBV cirrhosis, abstinence from alcohol in the alcoholic cirrhosis, immunosuppressive therapy in autoimmune cirrhosis.

CONTACTS AND LOCATIONS:
Overall Officials: Meropi D. Kontogianni, PhD, Study Director — Harokopio University
Locations (1):
- Harokopio University, Kallithea, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Data will be available upon demand.